CLINICAL TRIAL: NCT04264247
Title: Is There Any Relationship Between First Trimester (11-14 Weeks of Pregnancy) Fetal Thymus Volume and Preeclampsia? Prospective Cohort Study.
Brief Title: First Trimester Fetal Thymus Volume May Predict Preeclampsia
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ozlem Ece BASARAN, research assistant, Karadeniz Technical University
Other Study IDs: 2016/176
Record Dates: First submitted 2019-03-25; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2019-03

CONDITIONS: Preeclampsia
Keywords: Fetal thymus volume; Preeclampsia; Screening; Prediction
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Diagnostic Test: routine fetal ultrasonography at 11-14 weeks — routine fetal ultrasonography at 11-14 weeks

SUMMARY:
The exact etiology of preeclampsia remains unclear but is known to involve immunological factors. The thymus is one of the main organs involved in the development of the fetal immune system. The aim of this study was to explore the association between fetal thymus volume on ultrasound and preeclampsia by adding the 3-dimensional measurement of thymus volume to the routine fetal ultrasound scan at 11-14 week of gestation.

Investigators performed a prospective clinical study in 100 pregnant women in their first trimester of pregnancy who attended the Fetal Medicine Unit of the Medicine Faculty of Karadeniz Technical University during the study period. Maternal age, gravida, para, BMI, blood pressure, gestational age, CRL and fetal timus volume measured with VOCAL programme are recorded. For all patients routine clinical and ultrasound examinations were performed during pregnancy. Gestational age at birth, way of birth and newborn birthweight were recorded. The results were statistically compared in the SPSS 13.0 program. Student-t test and chi-square test were used for statistical analysis. ROC curve analysis was used for limit values. The data of patients with preeclampsia and without preeclampsia were compared. The ability of the thymus volume to predict the preeclampsia was tested using binary logistic regression analysis. P value <0.05 was considered statistically significant.

DETAILED DESCRIPTION:
The exact etiology of preeclampsia remains unclear but is known to involve immunological factors. The thymus is one of the main organs involved in the development of the fetal immune system. The aim of this study was to explore the association between fetal thymus volume on ultrasound and preeclampsia by adding the 3-dimensional measurement of thymus volume to the routine fetal ultrasound scan at 11-14 week of gestation.

ELIGIBILITY:
Inclusion Criteria:

* 11-14 weeks pregnancy with no abnormal ultrasonography evidence.

Exclusion Criteria:

Any history of obstetric complications Chronic hypertension Diabetes mellitus Infectious or autoimmune disease.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnancy
Study Population: 100 pregnancy women at 11-14 week of gestation were included in the study in the Obstetrics Department of Obstetrics and Gynecology of Medicine Faculty of Karadeniz Technical University, Medical Faculty of Medicine.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Preeclampsia | At least after 10 weeks of initial examination.
  Hypertension (Sistolik blood pressure >140, diastolic blood pressure >90), Proteinuria (>0.3 g proteinuria in 24 hour collected urine sample)

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem E Basaran, Principal Investigator — Karadeniz technical universty
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohamed N, Eviston DP, Quinton AE, Benzie RJ, Kirby AC, Peek MJ, Nanan RK. Smaller fetal thymuses in pre-eclampsia: a prospective cross-sectional study. Ultrasound Obstet Gynecol. 2011 Apr;37(4):410-5. doi: 10.1002/uog.8953. Epub 2011 Mar 7. PMID 21308839